CLINICAL TRIAL: NCT06901245
Title: The Effects of Tirzepatide in Young Adults With Prader-Willi Syndrome, Hypothalamic Obesity and General Non-Syndromic Obesity
Brief Title: Tirzepatide in PWS, HO and GNSO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Grace Kim (Other)
Collaborators: Vanderbilt University Medical Center (Other); Children's Hospitals and Clinics of Minnesota (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Grace Kim, Principal Investigator, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004995; I8F-NS-I001 (Other Grant/Funding Number: Lilly USA)
Record Dates: First submitted 2025-03-14; First posted 2025-03-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-01

CONDITIONS: Prader-Willi Syndrome; Hypothalamic Obesity; Obesity/Therapy
Keywords: Tirzepatide; GLP1 Agonist; Obesity; Prader-Willi Syndrome; Hypothalamic Obesity; General Obesity
MeSH Terms: conditions — Prader-Willi Syndrome; Sexual Infantilism; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Prader-Willi Syndrome (Active Comparator): Individuals 18-26 years with a BMI in the obesity range (BMI ≥95th percentile for age and sex or ≥30 kg/m2) with genetically confirmed Prader-Willi Syndrome between 18-26 years old.
  Interventions: Drug: Tirzepatide
- Hypothalamic Obesity (Active Comparator): Individuals 18-26 years with a BMI in the obesity range (BMI ≥95th percentile for age and sex or ≥30 kg/m2) and hypothalamic obesity as defined by damage to the medial hypothalamic region resulting in dysregulation of satiety and energy balance as diagnosed by a physician.
  Interventions: Drug: Tirzepatide
- General Non-Syndromic Obesity (Active Comparator): Individuals 18-26 years with a BMI in the obesity range (BMI ≥95th percentile for age and sex or ≥30 kg/m2) and general obesity unrelated to a genetic syndrome or underlying medical condition.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Subjects will take Tirzepatide for 48 weeks

SUMMARY:
This research study is comparing the effectiveness of a weight loss medication called Tirzepatide in young adults with Prader-Willi Syndrome and/or hypothalamic obesity, as compared to young adults with obesity that is unrelated to a genetic syndrome or underlying medical cause. These groups will be given medication for 1 year to see how weight and other health factors are effected by the medication.

DETAILED DESCRIPTION:
This study is for the following individuals:

* Age 18-26.
* Have Prader-Willi Syndrome, Hypothalamic Obesity, or Obesity unrelated to a genetic syndrome or medical condition.
* Have a BMI in the obesity range

If you/your child decide to take part in the research study, you/your child would participate in the study for approximately 56-60 weeks. During this time the following can be expected:

* Receive tirzepatide for once-weekly dosing.
* Complete 6 in-person SCH study visits
* Complete 4 telehealth visits.
* Complete the following research procedures:

  * Medical Record Review
  * Vital Signs
  * Anthropometry (e.g., height, weight, waist measurements)
  * Physical Exams
  * Laboratory Tests (e.g., fasting blood draws, urine test)
  * Dual-Energy Absorptiometry (DXA) scans
  * Questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18-26 years with a BMI in the obesity range (BMI ≥95th percentile for age and sex or ≥30 kg/m2) with either 1) genetically confirmed diagnosis of PWS, 2) hypothalamic obesity as defined by damage to the medial hypothalamic region resulting in dysregulation of satiety and energy balance as diagnosed by a physician, 3) general obesity unrelated to a genetic syndrome or underlying medical condition
* In a stable care setting at least 6 months prior to enrollment
* Able and willing to participate in study visits including tolerating blood draws, urine samples and tolerate DXA scan.
* Ability to take weekly subcutaneous tirzepatide
* Consistent caregiver if they are not independent
* Stable diet and exercise regimen for at least 6 months prior to enrollment
* Able to use contraceptive methods if able to conceive offspring in order to prevent unintentional pregnancy during the study

Exclusion Criteria:

* Current or recent (within 3 months of start of study drug initiation) use of weight loss medications
* Current use of insulin or sulfonylurea or other medication affecting insulin secretion or GLP1 clearance
* Current or prior use of any GLP1A or DPP4 inhibitor during the 6 months before screening
* Any medications that may affect the study endpoints
* Significant weight change (>3% weight gain or loss) in the last 2 months prior to enrollment
* Change in dose of chronic endocrine medications (testosterone, estrogen, levothyroxine, or growth hormone medications) >10%/kg/day for at least 3 months prior to study
* Current pregnancy or desire to become pregnant within study period, current lactation
* History of recurrent pancreatitis, CKD, gastroparesis
* Chronic/acute heart, kidney, or liver disease
* Personal or family history of medullary thyroid carcinoma or MEN syndrome type 2
* Uncontrolled diabetes (A1C >8.5%)
* DVT
* Cancer within the previous 5 years
* Current participation in an interventional clinical study
* Previous or planned surgical treatment for obesity
* Individuals with current substance abuse equivalnt to moderate or severe based on DSM 5 criteria (Hasin DS, 2013)
* Any suicidal ideation in the past year
* Unable to perform any of the procedures for the study
* Have a body weight, height, and/or width that that prohibits the ability to obtain accurate measurements according to the DXA manufacturer's specification
* Any condition that would prevent successful participation in the study.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 48 weeks
  Weight will be measured in kilograms through anthropometric measurements. Change in percent weight from baseline to week 48 of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity will then be assessed.

SECONDARY OUTCOMES:
Change in BMI | 48 weeks
  Change in BMI from baseline to 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity through anthropometric measurements. BMI will be calculated using weight (kg) and height (m) which will be combined to report BMI in kg/m^2. The percent change in this BMI value from baseline to 48 weeks will be calculated.
Change in fat mass | 48 weeks
  Change in fat mass (measured in kg by DXA scan) from baseline to 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity.
Change in appetite - CoEQ (Control of Eating Questionnaire) | 48 weeks
  Change in appetite during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity using an appetite questionnaire (CoEQ - Control of Eating Questionnaire). CoEQ is a 21-item scale to assess the severity and type of food cravings an individual experiences using a visual analog scale. Higher scores indicate higher severity of hyperphagia.
Change in appetite - Physician Rated Hyperphagia Severity Scale | 48 weeks
  Change in appetite during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity assed with a physician rated hyperphagia severity scale. This is a 5 point scale (0 to 5) to rate clinical imppression of hyperphagia severity. Higher scores mean more severity.
Change in metabolic markers - fasting lipids | 48 weeks
  Change in metabolic markers during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity including: fasting lipids via lipid profile assay via blood sample
Change in metabolic markers - fasting plasma glucose | 48 weeks
  Change in metabolic markers during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity including: fasting plasma glucose, via chemistry panel via blood sample
Change in metabolic markers- fasting insulin | 48 weeks
  Change in metabolic markers during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity including: fasting insulin via insulin assay via blood sample
Change in metabolic markers - hemoglobin A1C | 48 weeks
  Change in metabolic markers during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity including: hemoglobin A1C via hemoglobin A1C assay via blood sample
Change in metabolic markers- Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 48 weeks
  Change in metabolic markers during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity including: Homeostatic Model Assessment of Insulin Resistance (HOMA-IR). This is product measuring insulin resistance calculated using fasting insulin and fasting glucose values. Higher numbers indicate more insulins resistance.

OTHER OUTCOMES:
Change in safety markers -CBC | 48 weeks
  Change in safety markers during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity including: Complete Blood Count (CBC). This will be done with standard CBC assays via blood sample
Change in safety markers - CMP | 48 weeks
  Change in safety markers during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity including: Comprehensive Metabolic Panel (CMP). This will be done with standard CMP assays via blood sample.
Change in safety markers - coagulation factor assay PT [prothrombin time] | 48 weeks
  Change in safety markers during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity including: PT [prothrombin time], This assay will be done on drawn blood samples.
Change in safety markers - coagulation factor assay- PTT [Activated Partial Thromboplastin Time ] | 48 weeks
  Change in safety markers during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity including: , PTT [Activated Partial Thromboplastin Time ].This assay will be done on drawn blood samples.
Change in safety markers - coagulation factor assay - INR [international normalized ratio]. | 48 weeks
  Change in safety markers during 48 weeks of treatment with tirzepatide in young adults with PWS, HO, GNSO and obesity including: INR [international normalized ratio]. This assay will be done on drawn blood samples.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children's Minnesota, Saint Paul, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No